CLINICAL TRIAL: NCT02950753
Title: Does Intravenous Lactated Ringer Solution Raise Measured Serum Lactate?
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Medical Center of Southern Nevada (Other)
Responsible Party: Principal Investigator, Joseph (Tony) Zitek, MD, MD, University Medical Center of Southern Nevada
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: EM 2016.10
Record Dates: First submitted 2016-10-26; First posted 2016-11-01 (Estimated); Results first posted 2019-04-12 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-01

CONDITIONS: Hyperlactatemia
Keywords: Elevated Serum Lactate; Serum lactate; Ringer's Lactate; Lactated Ringer's; Hyperlactatemia
MeSH Terms: conditions — Hyperlactatemia | interventions — Ringer's Lactate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lactated Ringer (Experimental): Intravenous bolus of Lactated Ringer solution (30ml/kg) via 18ga IV catheter at wide open.
  Interventions: Drug: Lactated Ringer Solution
- Normal Saline (Placebo Comparator): Intravenous bolus of Normal Saline (30ml/kg) via 18ga IV catheter at wide open.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Lactated Ringer Solution — Fluid bolus of Lactated Ringer solution (30ml/kg).
  Other Names: LR
  Arms: Lactated Ringer
Drug: Normal Saline — Fluid bolus or Normal Saline (30ml/kg).
  Other Names: NS
  Arms: Normal Saline

SUMMARY:
Lactated Ringer's (LR) solution bolus is commonly administered in the emergency department setting to seriously ill patients. It is also common to obtain blood samples to determine serum lactate levels to aid in the assessment of the patient's degree of illness. This study endeavors to determine if serum lactate levels are affected by LR fluid administration in healthy adult individuals as compared to those who receive Normal Saline (NS). Healthy adult volunteers will be used as subjects so that the illness of hospital patients does not confound the results.

DETAILED DESCRIPTION:
Methods:

Approximately 30 subjects will be randomized to either the Lactated Ringer's group or the Placebo group. The study is powered to detect a difference of 0.3mmol/L between pre- and post-treatment lactate levels. All subjects are healthy volunteers over 18 years old. Healthy volunteers are defined as subjects with no acute symptoms who do not meet any of the exclusionary criteria below:

* Pregnancy or currently breast-feeding
* Prisoner status
* Those with any history of clinical conditions associated with fluid overload: congestive heart failure, renal, or hepatic failure
* Baseline serum lactate level >2.2mmol
* Baseline creatinine > 1.5 mg/dL

All volunteers will sign a written consent, approved by the Institutional Review Board (IRB). The consent form will discuss the risks and benefits of our study. The benefit of our study is to identify a possible confounder to our current interpretation of serum lactates. By clarifying whether Lactated Ringer's fluid can contribute to measured serum lactate level we hope to improve our care to septic patients and those patients with abnormal vital signs and elevated serum lactate levels in whom the diagnosis of sepsis is being considered. The risks of this study include the possible development of fluid overload state and pulmonary edema. We believe these sequelae would be very unlikely to occur since we are excluding anyone with a history of any clinical conditions associated with fluid overload.

The intended pool of our volunteer subjects will be from residents, attendings, hospital staff, and medical students in the hospital. Only healthy volunteers (as described previously) will be allowed to participate. Volunteer subjects from the hospital will be instructed to only participate after their work shifts or on their days off from work so as not to interfere with their job duties. The consent form will clearly specify that their participation in the study will not impact their academic status or employment. The subjects will also fill out a short data collection form that will have age, gender, known medical problems, medications, and allergies. The subjects will designate their weight in this consent form.

All subjects will receive an 18-gauge IV in one antecubital fossa. A second IV will be placed on the contralateral arm from which to draw serum studies.

The subjects randomized to the Lactated Ringer's arm will receive 30ml/kg Lactated Ringer's solution run wide open. Those randomized to the Placebo group will receive 30ml/kg of normal saline wide open. The precise fluid bolus quantity will be determined using a measure of the patient's weight in kilograms multiplied by 30, rounding the final figure to the nearest 100ml for simplicity. (E.g. 2077 ml would be rounded to 2100ml.) The pharmacist for the study will randomly assign each subject to a treatment group ensuring that there are an equal number of subjects in the Lactated Ringer's arm and in the Placebo arm. The pharmacist will obscure the fluid bag contents from the investigators to maintain the blinding. Only the pharmacist will know which treatment each subject received. The person administering the medications and those doing the analysis of the data will only know the study number of each patient, and will be blind to the pharmacist's randomization.

We have chosen a bolus of 30ml/kg Lactated Ringer's solution over one hour as the regimen for two reasons primarily. The first is that in a clinical scenario of sepsis or septic shock a 30ml/kg bolus is typical.[2] Therefore this protocol simulates what actually happens during the care of a septic patient. A second reason for the selection of a substantial quantity of LR given over a short time interval is to ensure detection of any change in serum lactate concentration secondary to this fluid bolus, if there is one to be found. A smaller quantity of LR over a shorter time span may result in a false negative result.

A serum lactate level will be drawn just prior to initiating treatment. Any subject found to have an abnormally high baseline serum lactate level (>2.2 mmol/L) before treatment will be excluded from the study.

The lactate will then be measured five minutes after the conclusion of the intravenous fluid treatment. 5ml of blood will be wasted to clear the line prior to this blood draw. Lactate will be measured with a point-of-care meter (the iSTAT-1 analyzer). The before-treatment and after-treatment lactate levels will be compared to see if the Lactated Ringer's caused a significant rise (>0.3 mmol/L) in the lactate level at any point during the data collection period.

The study design described previously lends itself to a brief investigation into an important clinical phenomenon during fluid resuscitation that will be investigated as a secondary outcome to this study. One consideration for the use of the Lactated Ringer's solution clinically is the incidence of hyperchloremic metabolic acidosis with the use of normal saline during fluid resuscitation.[8] Using our point-of-care meter (the iSTAT 1 analyzer) we will measure not only serum lactate but also a complete metabolic panel prior to and subsequent to the delivery of the 30 ml/kg fluid administration. We will subsequently analyze changes in serum sodium, chloride, potassium, and bicarbonate in each of the treatment groups, assessing for the degree of derangement that occurs in those electrolytes, and specifically evaluating for any trend toward hyperchloremic metabolic acidosis in the normal saline group.

While patients are in the process of receiving IV fluids, they will be kept on continuous cardiac and oxygenation monitoring. We believe it is highly unlikely that any subject will need any medical care during this study. However, let it be noted that there will be an attending and/or resident physician present at all times while patients are receiving treatment. Should any subject develop adverse effects as a result of our study, the physician will assess the patient and offer to register them in the emergency department. Any Serious Adverse Event (SAE) will be reported to the IRB within 5 days.

In order to protect the privacy of the research subjects and to maintain the confidentiality of the data, all data will be handled only by research assistants or investigators and will be stored in secure cabinets and on password protected computer files in the locked research offices. All research assistants and investigators are HIPAA-trained and credentialed by UMC IRB.

We have chosen a goal sample size of 30 based on the following calculation. A sample size of 25 achieves 80% power to detect a mean of paired differences of 0.3 with a known standard deviation of differences of 0.5 and with a significance level (alpha) or 0.05 using a one-sided paired t-test. To allow for patient drop out or equipment failure, we will aim to enroll 30 patients.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers
* 18 years and older

Exclusion Criteria:

* Pregnancy or currently breast-feeding
* Prisoner
* History of conditions associated with fluid overload: heart, renal or hepatic failure
* Baseline serum lactate level >2.2mmol
* Baseline creatinine > 1.5 mg/dL

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01-04 (Actual); Primary Completion 2017-05-05 (Actual); Study Completion 2017-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Zitek, MD, Principal Investigator — University Medical Center of Southern Nevada
Locations (1):
- University Medical Center of Southern Nevada, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
Identifiable Patient Data (IPD) will not be shared

REFERENCES:
- [Background] Zitek T, Cleveland N, Rahbar A, Parker J, Lim C, Elsbecker S, Forred W, Slattery DE. Effect of Nebulized Albuterol on Serum Lactate and Potassium in Healthy Subjects. Acad Emerg Med. 2016 Jun;23(6):718-21. doi: 10.1111/acem.12937. Epub 2016 May 11. PMID 26857949
- [Background] Kellum JA. Fluid resuscitation and hyperchloremic acidosis in experimental sepsis: improved short-term survival and acid-base balance with Hextend compared with saline. Crit Care Med. 2002 Feb;30(2):300-5. doi: 10.1097/00003246-200202000-00006. PMID 11889298
- [Result] Rivers E, Nguyen B, Havstad S, Ressler J, Muzzin A, Knoblich B, Peterson E, Tomlanovich M; Early Goal-Directed Therapy Collaborative Group. Early goal-directed therapy in the treatment of severe sepsis and septic shock. N Engl J Med. 2001 Nov 8;345(19):1368-77. doi: 10.1056/NEJMoa010307. PMID 11794169
- [Result] Dellinger RP, Levy MM, Rhodes A, Annane D, Gerlach H, Opal SM, Sevransky JE, Sprung CL, Douglas IS, Jaeschke R, Osborn TM, Nunnally ME, Townsend SR, Reinhart K, Kleinpell RM, Angus DC, Deutschman CS, Machado FR, Rubenfeld GD, Webb SA, Beale RJ, Vincent JL, Moreno R; Surviving Sepsis Campaign Guidelines Committee including the Pediatric Subgroup. Surviving sepsis campaign: international guidelines for management of severe sepsis and septic shock: 2012. Crit Care Med. 2013 Feb;41(2):580-637. doi: 10.1097/CCM.0b013e31827e83af. PMID 23353941
- [Result] ProCESS Investigators; Yealy DM, Kellum JA, Huang DT, Barnato AE, Weissfeld LA, Pike F, Terndrup T, Wang HE, Hou PC, LoVecchio F, Filbin MR, Shapiro NI, Angus DC. A randomized trial of protocol-based care for early septic shock. N Engl J Med. 2014 May 1;370(18):1683-93. doi: 10.1056/NEJMoa1401602. Epub 2014 Mar 18. PMID 24635773
- [Result] Mouncey PR, Osborn TM, Power GS, Harrison DA, Sadique MZ, Grieve RD, Jahan R, Harvey SE, Bell D, Bion JF, Coats TJ, Singer M, Young JD, Rowan KM; ProMISe Trial Investigators. Trial of early, goal-directed resuscitation for septic shock. N Engl J Med. 2015 Apr 2;372(14):1301-11. doi: 10.1056/NEJMoa1500896. Epub 2015 Mar 17. PMID 25776532
- [Result] ARISE Investigators; ANZICS Clinical Trials Group; Peake SL, Delaney A, Bailey M, Bellomo R, Cameron PA, Cooper DJ, Higgins AM, Holdgate A, Howe BD, Webb SA, Williams P. Goal-directed resuscitation for patients with early septic shock. N Engl J Med. 2014 Oct 16;371(16):1496-506. doi: 10.1056/NEJMoa1404380. Epub 2014 Oct 1. PMID 25272316
- [Result] Didwania A, Miller J, Kassel D, Jackson EV Jr, Chernow B. Effect of intravenous lactated Ringer's solution infusion on the circulating lactate concentration: Part 3. Results of a prospective, randomized, double-blind, placebo-controlled trial. Crit Care Med. 1997 Nov;25(11):1851-4. doi: 10.1097/00003246-199711000-00024. PMID 9366769

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lactated Ringer | Normal Saline
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lactated Ringer | Normal Saline | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 8 | 11
  Male | 12 | 7 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Lactate Level of the LR Group Compared to the NS Group.
Description: Final mean lactate minus initial mean lactate
Time Frame: 5 minutes after IV bolus has ended.
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Lactated Ringer | Normal Saline
Number analyzed (Participants) | 15 | 15
mmol/L | 0.93 [0.42 to 1.44] | 0.37 [-0.26 to 1.00]

2. Secondary Outcome: Decrease in Bicarbonate Level of the LR Group Compared to the NS Group
Description: Baseline serum bicarbonate will be measured in both groups just prior to IV administration and again at 5 minutes after IV bolus has ended.
Time Frame: 5 minutes after IV bolus has ended.
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Lactated Ringer | Normal Saline
Number analyzed (Participants) | 15 | 15
mEq/L | -0.36 (2.6) | 2.35 (2.1)

3. Secondary Outcome: Final Chloride Level Minus Initial Chloride Level of the LR Group Compared to the NS Group
Description: Baseline serum chloride will be measured in both groups just prior to IV administration and again at 5 minutes after IV bolus has ended.
Time Frame: 5 minutes after IV bolus has ended.
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Lactated Ringer | Normal Saline
Number analyzed (Participants) | 15 | 15
mEq/L | -0.4 (2.4) | 3.7 (1.4)

ADVERSE EVENTS:
Time Frame: Subjects were monitored for adverse events during the study period and for five minutes afterward (total of about one hour).
Arm/Group | Lactated Ringer | Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-17): https://cdn.clinicaltrials.gov/large-docs/53/NCT02950753/Prot_SAP_000.pdf